CLINICAL TRIAL: NCT02173444
Title: Comparison of the Accuracy and Reliability of AMH, FSH and AFC in Predicting Ovarian Response
Acronym: AMH FSH AFC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vietnam National University (Other)
Responsible Party: Principal Investigator, Manh Tuong Ho, Doctor, Vietnam National University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1234-DHYD
Record Dates: First submitted 2014-06-23; First posted 2014-06-25 (Estimated); Last update posted 2014-06-25 (Estimated); Status verified 2014-06

CONDITIONS: Infertility
Keywords: in-vitro fertilization; ovarian stimulation
MeSH Terms: conditions — Infertility | interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Blood test

SUMMARY:
Serum bio-markers have different prediction values for ovarian response during ovarian stimulation in-vitro fertilization

ELIGIBILITY:
Inclusion Criteria:

* Age ≤ 45 years at the time of FSH starting
* BMI < 25 kg/m2,
* First IVF attempt
* Receiving GnRH-antagonist protocol
* Had oocyte retrieval

Exclusion Criteria:

* Had ovarian stimulation or ovulation induction within 2 months prior to the study
* PCOS
* Had ovarian tumor or endometrioma
* Hyperprolactinemia
* Thyroid hormone disorders
* Pituitary failure
* Had other medical situations such as liver failure, renal failure, heart disease, diabetes, depression
* Had IVM

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 820 (Actual)
Dates: Start 2013-01; Primary Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Number of oocytes | At the time of oocyte retrieval
number of oocytes at time of oocyte retrieval | up to 14 days

CONTACTS AND LOCATIONS:
Locations (1):
- An Sinh Hospital, Ho Chi Minh City, Ho Chi Minh, Vietnam